CLINICAL TRIAL: NCT07055633
Title: Improving Cognitive Rehabilitation Outcomes for Veterans With mTBI+PTSD
Brief Title: Improving Cognitive Rehabilitation Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRD1-012-24W; RRD1-012-24W (Other Grant/Funding Number: VA Rehabilitation Research Development and Transla)
Record Dates: First submitted 2025-06-24; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Mild Traumatic Brain Injury; Posttraumatic Stress Disorder
Keywords: brain injury; posttraumatic stress disorder
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic; Brain Injuries

STUDY DESIGN:
Intervention Model Description: CCT+MBLT vs CCT+ION
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CCT+MBLT (Experimental): Compensatory Cognitive Training + Morning Bright Light Therapy
  Interventions: Device: CCT+MBLT
- CCT+ION (Sham Comparator): Compensatory Cognitive Training + Negative Ion Generator
  Interventions: Device: CCT+ION

INTERVENTIONS:
Device: CCT+MBLT — Compensatory Cognitive Training + Morning Bright Light Therapy (Aurora LightPad)
  Other Names: Morning Bright Light Therapy Aurora LightPad lightbox
  Arms: CCT+MBLT
Device: CCT+ION — Compensatory Cognitive Training + Negative Ion Generator (SphereOne)
  Other Names: SphereOne negative ion generator
  Arms: CCT+ION

SUMMARY:
Posttraumatic stress disorder (PTSD) and mild TBI (mTBI) frequently co-occur in post-9/11 Veterans, and together are associated with worse cognitive performance, mental health, everyday functioning, community integration, quality of life, and treatment response than either condition alone. Additional comorbidities, such as depression and sleep disturbance, are common and further exacerbate these problems. The investigators will investigate Compensatory Cognitive Training (CCT) and Morning Bright Light Therapy (MBLT) vs Negative Ion Generator (ION), to directly target cognition, depression, and sleep disturbance and to improve CCT-associated rehabilitation outcomes. The investigator's randomized controlled trial in 144 Veterans with mTBI+PTSD across two VA sites will compare cognition, functioning, and other secondary outcomes following CCT+MBLT vs. CCT+ION. This study addresses the significant gap in services and evidence-based treatments for Veterans with mTBI+PTSD.

DETAILED DESCRIPTION:
The investigators aim to compare CCT+MBLT with CCT+ION for improving cognition, functioning, and secondary outcomes in Veterans with mTBI+PTSD.

Objective cognitive performance and everyday functioning are co-primary outcomes. Depression and sleep disturbance are target mechanisms and secondary outcomes include PTSD symptom severity, post-concussive symptom severity, cognitive symptom severity, and quality of life.

Improvements in mood and sleep will be investigated as mediators. To explore for whom these interventions are most effective, the investigators will evaluate whether individual difference variables (e.g., demographics, premorbid functioning, treatment adherence) or baseline performance on primary and secondary outcome measures moderate intervention-related improvements in objective cognitive performance and everyday functioning.

The investigators will enroll a representative sample of 144 post-9/11 Veterans with mTBI+PTSD at two VA sites (San Diego and Portland). Assessments will be conducted at baseline, mid-treatment (5 weeks), post-treatment (10 weeks), and three-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Post 9/11 Veterans enrolled at VA San Diego or VA Portland
* Ability to provide informed consent
* Living independently
* History of mTBI confirmed by OSU-TBI
* Current diagnosis of PTSD confirmed by CAPS-5
* Current cognitive concerns ("Do you have concerns about your cognition, thinking, attention, or memory?")
* Current concern regarding depression and/or sleep disturbance; defined by a score of 5 on the PHQ-9 and/or 8 on the ISI, respectively (score of 2 or higher on ISI item 1, 2, or 3, reflecting at least "moderate" difficulty with falling asleep, staying asleep, or waking up too early in the morning)

Exclusion Criteria:

* Current substance use disorder with <30 days abstinence
* History of primary psychotic disorder
* History of moderate to severe TBI (loss of consciousness >30 minutes)
* History of macular degeneration or bipolar disorder (both contraindicated for bright light therapy)
* Not work night or swing shift schedules
* Untreated obstructive sleep apnea either via self-report or a score 5 on the STOP-BANG
* Current engagement in bright light therapy
* Auditory or visual impairments precluding participation in assessments or treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Cognitive Performance | baseline, 10 weeks
  Composite z score of Hopkins Verbal Learning Test-Revised; Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) Digit Span; WAIS-IV Coding; Delis-Kaplan Executive Function System (D-KEFS) Trails; D-KEFS Color-Word Interference; and the UCSD Performance-Based Skills Assessment-Brief (UPSA-B). There is no minimum or maximum value of a z score. Higher scores will reflect better outcomes.
Functioning | baseline, 10 weeks
  Composite z score of Brief Inventory of Psychosocial Functioning and the World Health Organization Disability Assessment Schedule 2.0. There is no minimum or maximum value of a z score. Higher scores will reflect better outcomes.

SECONDARY OUTCOMES:
Insomnia Severity Index | baseline, 10 weeks
  Insomnia severity. Scores range from 0-28, with higher scores representing worse insomnia.
Pittsburgh Sleep Quality Index | baseline, 10 weeks
  Sleep quality. Scores range from 0-21, with higher scores representing worse sleep quality.
Total Sleep Time | baseline, 10 weeks
  Total Sleep Time derived from Actiwatch2. Minutes range from 0 to 1440 per day, with higher numbers reflecting more minutes of sleep.
Patient Health Questionnaire-9 | baseline, 10 weeks
  Depression symptom severity. Scores range from 0-27, with higher scores reflecting worse depression symptoms.
PTSD Checklist for DSM-5 | baseline, 10 weeks
  PTSD symptom severity. Scores range from 0-80, with higher scores reflecting worse PTSD symptoms.
Neurobehavioral Symptom Inventory | baseline, 10 weeks
  Postconcussive symptom severity. Scores range from 0-88, with higher scores reflecting worse neurobehavioral symptoms.
Subjective cognitive functioning | baseline, 10 weeks
  Mean score across Neuro-QOL Applied Cognition Executive Function and Neuro-QOL Applied Cognition General Concerns scales. The mean score has a range of 8-40, with higher scores reflecting better subjective cognitive functioning.
World Health Organization Quality of Life | baseline, 10 weeks
  Quality of life. Scores range from 0-100, with higher scores reflecting better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth W. Twamley, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (2):
- United States (2):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Portland Health Care System, Portland, OR, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No